CLINICAL TRIAL: NCT05861973
Title: SMARTer Weight Loss Management
Acronym: SMARTer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Florida State University (Other)
Responsible Party: Principal Investigator, Bonnie Spring, Krafft Professor of Behavioral Sciences and Social Medicine and Director of Florida Blue Center for Rural Health Research & Policy, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00005828
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: stepped care; adaptive intervention; non-inferiority trial; behavioral obesity treatment
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This is a randomized control trial with 3 parallel intervention arms. One arm will be the SMARTer active treatment group, one the active DPP treatment group, and the other a Self-Guided control group. Assessors will be blinded to study condition, and intervention will be behavioral.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adaptive SMARTer intervention (SMARTer) (Experimental): Smartphone application, diet and activity goals, online lessons, brief remote sessions with a Health Promotionist. Data from a wifi scale will be monitored. Individuals losing less than .5 lb per week will be stepped up to also be given meal replacement products. Will have physical measures taken at baseline, 3 months, 6 months, 9 months, and 12 months.
  Interventions: Behavioral: Adaptive SMARTer intervention (SMARTer)
- Diabetes Prevention Program (DPP) (Experimental): Fixed intervention using participant program manual, diet and activity logs, hour long remote sessions with a Health Promotionist. Will have physical measures taken at baseline, 3 months, 6 months, 9 months, and 12 months.
  Interventions: Behavioral: Diabetes Prevention Program (DPP)
- Self-Guided Treatment (Self-Guided) (Active Comparator): Provides paper and internet resources tailored to geographic area, educating on leading a healthier lifestyle, including information on wellness and physical activity. Will have physical measures taken at baseline, 3 months, 6 months, 9 months, and 12 months.
  Interventions: Behavioral: Self-Guided Treatment (Self-Guided)

INTERVENTIONS:
Behavioral: Adaptive SMARTer intervention (SMARTer) — Participants will receive calorie, fat, and physical activity goals, a Smartphone application for self-monitoring their diet, activity and weight, online educational readings, and brief bi-weekly remote health sessions with a Health Promotionist. They will also be loaned a Fitbit tracking device and a wireless Bluetooth scale for 12 months.
  Arms: Adaptive SMARTer intervention (SMARTer)
Behavioral: Diabetes Prevention Program (DPP) — In accordance with the Center for Disease Control curriculum, participants will receive a participant log for tracking physical activity, food intake, and weight, a paper participant guide with worksheets, logs, and psycho-educational materials, and 16 hour long remote sessions with a Health Promotionist.
  Arms: Diabetes Prevention Program (DPP)
Behavioral: Self-Guided Treatment (Self-Guided) — Provides paper and internet resources tailored to geographic area, educating on leading a healthier lifestyle, including information on wellness and physical activity. Will have physical measures taken at baseline, 3 months, 6 months, 9 months, and 12 months.
  Arms: Self-Guided Treatment (Self-Guided)

SUMMARY:
The SMARTer trial will be a three-arm, randomized controlled non-inferiority trial that compares the optimized, adaptive SMARTer intervention, fixed DPP, and Self-Guided (Control). The trial will address whether a scalable, stepped-care intervention can stand up to gold-standard DPP by achieving comparable weight loss at a lower cost. Alongside evaluation of clinical non-inferiority, a comprehensive economic evaluation will inform relative affordability. Cost information is important to inform treatment policy and change standard of care, but is sorely lacking for behavioral interventions. The SMARTer intervention reduces costs by initially offering minimal intervention to all and stepping up to offer more costly treatment components only to non-responders who fail to attain the target weight loss. A rigorous economic evaluation planned and designed alongside the SMARTer trial will provide an accurate, robust head-to-head comparison of costs, cost-effectiveness, and projected lifetime health care costs between the three arms.

DETAILED DESCRIPTION:
The proposed study seeks to test the hypothesis that SMARTer is non-inferior to DPP in its effect on 6-month weight loss. During the 24-week active intervention phase, participants will be randomized to one of three first-line treatments: 1) the adaptive SMARTer intervention, 2) fixed DPP, or 3) usual care assessment-only (control). Participants will be assessed at 3-month, 6-month, 9-month, and 12-month timepoints to evaluate overall weight loss, and to explore whether SMARTer is cost-effective compared to DPP or standard care.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* BMI of ≥25, weight <396 lbs
* Must own a Smartphone, and be willing to install the SMARTer app
* Not enrolled in a formal weight loss program

Exclusion Criteria:

* Cerebrovascular accident or myocardial infarction within six months of enrollment
* Diabetes treated with insulin
* Pregnancy, lactation or intended pregnancy
* Active suicidal ideation
* Anorexia or bulimia
* Requiring an assistive device for mobility
* Taking weight loss medications, such as GLP-1 agonists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Weight | Baseline to 6-Months
  Participant change in weight, in pounds, from baseline to 6-months.

SECONDARY OUTCOMES:
Cost | 12 Months
  Costs of SMARTer versus DPP versus Control implementation. We will utilize a micro-costing approach to capture all costs associated with the implementation of the treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Spring, PhD, Principal Investigator — Florida State University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No